CLINICAL TRIAL: NCT03325686
Title: Efficacy of Vitamin D Supplementation in Physical Performance of Iranian Elite Athletes
Brief Title: Vitamin D Supplementation in Physical Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Tirang R. Neyestani, Ph.D., Professor, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 054-575
Record Dates: First submitted 2017-10-20; First posted 2017-10-30 (Actual); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Healthy; Athletes
Keywords: vitamin D; atletes; physical performance
MeSH Terms: interventions — Fumigant 93

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vitamin D supplement (Experimental): D
  Interventions: Dietary Supplement: vitamin D supplement
- control (Placebo Comparator): P
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: vitamin D supplement — D; received 50,000 IU of vitamin D supplement weekly
  Other Names: D
  Arms: vitamin D supplement
Other: Placebo — placebo
  Other Names: P
  Arms: control

SUMMARY:
This study was performed to evaluate the efficacy of weekly vitamin D supplementation on athletic performance in Iranian athletes

DETAILED DESCRIPTION:
Seventy subjects were enrolled in the study. The athletes were randomly divided into two groups: vitamin D supplement (D; received 50,000 IU of vitamin D supplement weekly) and control (P, received a placebo weekly). Duration of the study was eight weeks. Anthropometric, dietary, athletic performance and biochemical evaluations were performed for all subjects in the beginning and in the end of the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* professional athletes

Exclusion Criteria:

* receiving vitamin D supplement in past 3 months

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Changes from baseline serum 25-hydroxy vitamin D at eight weeks | 8 weeks
  nmol/L

SECONDARY OUTCOMES:
Changes from baseline Truncal Fat at eight weeks | 8 weeks
  percent
Changes from baseline visceral fat at eight weeks | 8 weeks
  percent
Changes from Strength leg press at 8 weeks | 8 weeks
  percent
Changes from Ergojump at 8 weeks | 8 weeks
  percent
Changes from baseline Vertical jump at 8 weeks | 8 weeks
  percent
Change from baseline Agility at 8 weeks | 8 weeks
  percent
changes from Speed at 8 weeks | 8 weeks
  percent

CONTACTS AND LOCATIONS:
Overall Officials: Tirang R. Neyestani, PhD, Study Chair — Laboratory of Nutrition Research, National Nutrition and Food Technology Research Institute (NNFTRI) and Faculty of Nutrition Science and Food Technology, Shahid Beheshti University of Medical Sciences, Tehran, Iran
Locations (1):
- National Nutrition and Food Technology Research Institute, Tehrān, Tehran Province, Iran

IPD SHARING:
Plan to Share IPD: Undecided